CLINICAL TRIAL: NCT04565275
Title: A Multi-center Open-label, Phase I/II Clinical Trial to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of ICP-192 in Patients With Advanced Solid Tumors and FGFR Gene Alterations
Brief Title: A Study of ICP-192 in Patients With Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing InnoCare Pharma Tech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ICP-CL-00303
Record Dates: First submitted 2020-09-01; First posted 2020-09-25 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Advanced Solid Tumors; Urothelial Carcinoma; Cholangiocarcinoma
MeSH Terms: conditions — Carcinoma, Transitional Cell; Cholangiocarcinoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ICP-192 (Experimental): 1. Dose Escalation Phase ICP-192
  2. Dose Expansion Phase ICP-192
  Interventions: Drug: Drug ICP-192

INTERVENTIONS:
Drug: Drug ICP-192 — 1. Dose Escalation Phase ICP-192 will be taken by patients with advanced solid tumor and will be treated follow the "3+3" dose escalation scheme
  2. Dose Expansion Phase ICP-192 will be taken by patients with urothelial carcinoma or cholangiocarcinoma with FGFR gene alterations and will be treated at a single dose defined from the Dose Escalation Phase.

SUMMARY:
This is a multi-center, open-label, phase I/II clinical study to evaluate ICP-192 in patients with advanced solid tumors and FGFR gene alterations. It consists of two parts: Part I (Phase I), dose escalation and Part II (Phase II), dose expansion.

DETAILED DESCRIPTION:
Part I (Phase I) of the study enrolls patients with advanced solid tumors (9-15 patients); Part II (Phase II) of the study enrolls patients with urothelial carcinoma or cholangiocarcinoma with FGFR genetic alterations (30 patients).

ELIGIBILITY:
Major Inclusion Criteria

Participants are eligible to be included in the study only if all of the following criteria apply:

1. Participate voluntarily, sign informed consent, and follow the study treatment plan and scheduled visits;
2. Phase I: Patients with histologically or cytologically confirmed unresectable or metastatic advanced malignant solid tumors who have progressed under standard treatment or recurred after or were intolerant to all standard treatment regimens, or have no standard treatment available;
3. Phase II: patients with histologically or cytologically confirmed unresectable or metastatic urothelial carcinoma or cholangiocarcinoma, who have progressed or recurred after or were intolerant to first-line chemotherapy, or have progressed/relapsed within 12 months after neoadjuvant /adjuvant chemotherapy;
4. Phase II: Existing test reports have confirmed the FGFR gene alteration or the central laboratory has detected the FGFR gene alteration.
5. Age ≥18 years old;
6. At least one measurable lesion according to the Response Evaluation Criteria of Solid Tumor, version 1.1 (RECIST 1.1);
7. ECOG performance status of 0-1;
8. Life expectancy for more than 3 months; Must have adequate organ function Major Exclusion Criteria

Participants are excluded from the study if any of the following criteria apply:

1. Have previously been treated with selective pan-FGFR molecular inhibitors or antibody drugs, except for the FGFR4 selective inhibitors;
2. Within 2 weeks before the first dose of study drug, the subject's phosphate level continuing to exceed the ULN despite medical treatment;
3. Patients with clinically significant gastrointestinal dysfunction
4. Has known central nervous system metastases;
5. Has a history of or currently uncontrolled cardiovascular diseases
6. History of organ transplantation or a history of allogeneic hematopoietic stem cell transplantation;
7. Current evidence of corneal or retinal abnormalities that may increase eye toxicity;
8. Active hepatitis B virus active hepatitis C, or HIV infection;
9. Has not recovered from reversible toxicity of prior anti-tumor therapy
10. Pregnant or lactating women, as well as women with childbearing potential who are unwilling or unable to perform contraception from the screening to 6 months after the last study drug administration; and fertile men who are unwilling or unable to perform contraception from screening to 3months after the last study drug administration
11. Other conditions considered by the investigator to be inappropriate for participation in this study.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2023-11-30 (Estimated); Study Completion 2024-04-15 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | Up to 3 years
  Phase I: Dose Escalation & Phase II: Dose Expansion To evaluate the safety and tolerability of different doses of ICP-192 in patients with advanced solid tumors
MTD | Up to 3 years
  Phase I: Dose Escalation To determine Maximum Tolerated Dose（MTD) for ICP-192
OBD | Up to 3 years
  Phase I: Dose Escalation To determine Optimal Biological Dose (OBD) for ICP-192
RP2D | Up to 3 years
  Phase I: Dose Escalation To determine Recommended Phase 2 Dose (RP2D) for ICP-192
ORR | Up to 3 years
  Phase II: Dose Expansion Objective Response Rate

SECONDARY OUTCOMES:
Peak concentration (Cmax) | Up to 3 years
  Phase I: Dose Escalation Peak concentration (Cmax)
AUC | Up to 3 years
  Phase I: Dose Escalation AUC
DCR | Up to 3 years
  Phase II: Dose Expansion disease control rate
DOR | Up to 3 years
  Phase II: Dose Expansion duration of response
PFS | Up to 3 years
  Phase II: Dose Expansion progression-free survival
OS | Up to 3 years
  Phase II: Dose Expansion overall survival

OTHER OUTCOMES:
Drug exposure | Up to 3 years
  Phase II: Dose Expansion Assessment of the correlations between drug exposure (e.g., AUC, Cmax) and patient response to ICP-192.
PD biomarker | Up to 3 years
  Phase II: Dose Expansion Assessment of the correlations between PD biomarker and patient response to ICP-192.

CONTACTS AND LOCATIONS:
Locations (16):
- United States (9):
  - Arizona Oncology, Tucson, Arizona
  - University of California, San Diego (UCSD) - Moores Cancer Center, La Jolla, California
  - Rocky Mountain Cancer Centers, Aurora, Colorado
  - Mid Florida Hematology and Oncology, Orange City, Florida
  - Minnesota Oncology Hematology, Minneapolis, Minnesota
  - Clinical Research Alliance, Lake Success, New York
  - Rutgers Cancer Institute of New Jersey, The Bronx, New York
  - The Ohio State University, Columbus, Ohio
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
- Australia (7):
  - Macquarie University Hospital, Macquarie Park, New South Wales
  - GenesisCare - North Shore, St Leonards, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Pindara Private Hospital, Benowa, Queensland
  - Monash Medical Centre Clayton, Clayton, Victoria
  - Peninsula & South Eastern Haematology & Oncology Group, Frankston, Victoria
  - Olivia Newton-John Cancer Research Institute, Melbourne, Victoria